CLINICAL TRIAL: NCT02906488
Title: Special Drug Use Results Survey of Safety and Efficacy of Long-term (104 Weeks) Use of Duodopa Enteral Solution in Patients With Parkinson's Disease in Actual Usage Condition
Brief Title: Special Drug Use-results Survey of Duodopa Enteral Solution in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-720
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease
Keywords: Quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Parkinson's Disease

SUMMARY:
The purpose of this study is to assess the safety and efficacy of long-term use of Duodopa in patients with Parkinkon's disease in actual usage

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Parkinson's disease using Duodopa for the purpose of improving circadian change (wearing-off phenomenon) of symptoms of Parkinson's disease in which sufficient effect cannot be obtained with existing drug therapy including levodopa-containing drugs.

Exclusion Criteria:

NA

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease using Duodopa for the purpose of improving circadian change (wearing-off phenomenon) of symptoms of Parkinson's disease in which sufficient effect cannot be obtained with existing drug therapy including levodopa-containing drugs.
Sampling Method: Non-Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Change in "Off" Periods From Start of Treatment to Week 104 | 104 weeks
  "Off" periods describe those times when medication is not working well and a person has greater difficulty with movement.

SECONDARY OUTCOMES:
Time-dependent Change in "Off" Time and "On" Time Accompanied By Dyskinesia Interfering with Daily Activities | 104 Weeks
  "Off" periods describe those times when medication is not working well and a person has greater difficulty with movement, and "On" periods describe when medication is working well and symptoms are controlled.
Time-dependent Change in Unified Parkinson's Disease Rating Scale (UPDRS) | 104 Weeks
  Motor evaluation
Time-dependent Change in Parkinson's Disease Questionnaire - 8 Items (PDQ-8) | 104 weeks
  The PDQ-8 is a quality of life questionnaire for PD patient. This short-form version derived from the PDQ-39 includes 1 question from each of the domains on the PDQ-39 (mobility, ADLs, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort).
"Off" Period and "On" Period Accompanied by Dyskenesia Interfering with Daily Activities by Patient Characteristic Factor | 104 weeks
  "Off" periods describe those times when medication is not working well and a person has greater difficulty with movement, and "On" periods describe when medication is working well and symptoms are controlled.
Time-dependent Change in Parkinson's Disease Quality of Life Questionnaire - Carers (PDQ-Carer) | 104 weeks
  The PDQ-Carer is a 29 item measure of health related quality of life for use with carers of people with Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (127):
- Japan (127):
  - Nagoya University Hospital /ID# 212303, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 166893, Nagoya, Aichi-ken
  - Toyota Memorial Hospital /ID# 166891, Toyota-shi, Aichi-ken
  - Akita City Hospital /ID# 207121, Akita, Akita
  - National Hospital Organization Akita National Hospital /ID# 207374, Yurihonjo-shi, Akita
  - Aomori Prefectural Central Hospital /ID# 165286, Aomori, Aomori
  - Kameda General Hospital /ID# 166906, Kamogawa-shi, Chiba
  - Juntendo University Urayasu Hospital /ID# 162890, Urayasu-shi, Chiba
  - Saiseikai Matsuyama hospital /ID# 169561, Matsuyama, Ehime
  - Saiseikai Saijo Hospital /ID# 167705, Saijo-shi, Ehime
  - Ehime University Hospital /ID# 162889, Toon-shi, Ehime
  - Fukui Red Cross Hospital /ID# 166907, Fukui-shi, Fukui
  - Fukuoka University Hospital /ID# 166900, Fukuoka, Fukuoka
  - Kitakyushu Yahata Higashi Hospital /ID# 213849, Kitakyushu-shi, Fukuoka
  - Wakamatsu Hospital /ID# 160818, Kitakyusyu-shi, Fukuoka
  - Fukushima Medical University Hospital /ID# 169560, Fukushima, Fukushima
  - Gifu Municipal Hospital /ID# 207777, Gifu, Gifu
  - Gifu Prefectural General Medical Center /ID# 166894, Gifu, Gifu
  - Gifu University Hospital /ID# 207378, Gifu, Gifu
  - Mihara Memorial /ID# 252885, Isesaki-shi, Gunma
  - SUBARU Health Insurance Society Ota Memorial Hospital /ID# 207778, Ota-shi, Gunma
  - National Hospital Organization Takasaki General Medical Center /ID# 207773, Takasaki-shi, Gunma
  - Hiroshima City Hiroshima Citizens Hospital /ID# 207126, Hiroshima, Hiroshima
  - Hiroshima Teishin Hospital /ID# 245072, Hiroshima, Hiroshima
  - Hiroshima University Hospital /ID# 212269, Hiroshima, Hiroshima
  - Japanese Red Cross Asahikawa Hospital /ID# 207149, Asahikawa-shi, Hokkaido
  - National Hospital Organization Asahikawa Medical Center /ID# 155744, Asahikawa-shi, Hokkaido
  - Date Red Cross Hospital /ID# 207776, Date-shi, Hokkaido
  - Hakodate Municipal Hospital /ID# 212304, Hakodate-shi, Hokkaido
  - Muroran-Clinic /ID# 207780, Muroran-shi, Hokkaido
  - Obihiro kosei Hospital /ID# 166904, Obihiro-shi, Hokkaido
  - Hokuto Hospital /ID# 207850, Obihiro-shi, Hokkaido
  - Sapporo Medical University Hospital /ID# 207373, Sapporo, Hokkaido
  - Sapporo City General Hospital /ID# 212305, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 166902, Sapporo, Hokkaido
  - Hokkaido Medical Center /ID# 161763, Sapporo, Hokkaido
  - Sapporo Neurology Hospital /ID# 207779, Sapporo, Hokkaido
  - Himeji Central Hospital /ID# 164136, Himeji-shi, Hyōgo
  - Kobe Home Clinic of Neurology /ID# 212308, Kobe, Hyōgo
  - Kobe University Hospital /ID# 166895, Kobe, Hyōgo
  - Nishi-Kobe Medical Center /ID# 207781, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 169562, Nishinomiya-shi, Hyōgo
  - Hyogo-Chuo National Hospital /ID# 207376, Sanda-shi, Hyōgo
  - Hyogo College of Medicine Sasayama Medical Center /ID# 208716, Tanbasasayama-shi, Hyōgo
  - Toyooka Hospital /ID# 212270, Toyooka-shi, Hyōgo
  - Ryugasaki Saiseikai Hospital /ID# 207846, Ryugasaki-shi, Ibaraki
  - JA Toride Medical Center /ID# 212302, Toride-shi, Ibaraki
  - Iwate Medical University Uchimaru Medical Center /ID# 212265, Morioka, Iwate
  - Minami Kyushu National Hospital /ID# 171052, Aira-shi, Kagoshima-ken
  - Okatsu Hospital /ID# 213489, Kagoshima, Kagoshima-ken
  - Kagoshima University Hospital /ID# 166909, Kagoshima, Kagoshima-ken
  - Kikuno Hospital /ID# 207784, Minamikyusyu-shi, Kagoshima-ken
  - Tokai University Hospital /ID# 250954, Isehara, Kanagawa
  - St Marianna University School Of Medicine /ID# 204347, Kawasaki-shi, Kanagawa
  - St Marianna University School Of Medicine /ID# 207119, Kawasaki-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital /ID# 160825, Sagamihara-shi, Kanagawa
  - Yokohama City University Medical Center /ID# 165285, Yokohama, Kanagawa
  - Kochi Medical School Hospital /ID# 166903, Nankoku-shi, Kochi
  - Kumamoto Saishunso National Hospital /ID# 212813, Kōshi, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine /ID# 207130, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 162891, Kyoto, Kyoto
  - National Hospital Organization Utano National Hospital /ID# 164139, Kyoto, Kyoto
  - Mie University Hospital /ID# 164140, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 169557, Sendai, Miyagi
  - NHO Sendai Nishitaga National Hospital /ID# 164977, Sendai, Miyagi
  - Tohoku Medical and Pharmaceuti /ID# 169558, Sendai, Miyagi
  - National Hospital Organization Sendai Medical Center /ID# 160831, Sendai, Miyagi
  - Kobayashi City Hospital /ID# 208715, Kobayashi-shi, Miyazaki
  - Fujimoto General Hospital /ID# 207150, Miyakonojo-shi, Miyazaki
  - Ina Central Hospital /ID# 166905, Ina-shi, Nagano
  - Aizawa Hospital /ID# 212307, Matsumoto-shi, Nagano
  - Shinshu University Hospital /ID# 169559, Matsumoto-shi, Nagano
  - Nagasaki Kita Hospital /ID# 204353, Nishisonogi-gun, Nagasaki
  - Nara Medical University Hospital /ID# 160830, Kashihara-shi, Nara
  - Minami Nara General Medical Center /ID# 207372, Yoshino-gun, Nara
  - NHO Niigata National Hospital /ID# 204337, Kashiwazaki-shi, Niigata
  - Nagaoka Red Cross Hospital /ID# 212301, Nagaoka-shi, Niigata
  - Midori Hospital /ID# 207127, Niigata, Niigata
  - Oita Prefectural Hospital /ID# 208714, Ōita, Oita Prefecture
  - Japanese Red Cross Okayama Hospital /ID# 212268, Okayama, Okayama-ken
  - Okayama Kyokuto Hospital /ID# 166892, Okayama, Okayama-ken
  - Nanbu Medical Center / Nanbu Child Medical Center /ID# 207148, Shimajiri-gun, Okinawa
  - Higashiosaka City Medical Center /ID# 166901, Higashiosaka-shi, Osaka
  - Izumi City General Hospital /ID# 207775, Izumi-shi, Osaka
  - Kayashimaikuno Hospital /ID# 171051, Kadoma-shi, Osaka
  - Mino City Hospital /ID# 161765, Minoh, Osaka
  - Osaka Saiseikai Nakatsu Hospital /ID# 168357, Osaka, Osaka
  - Kitano Hospital, Tazuke Kofukai Medical Research Institute /ID# 259507, Osaka, Osaka
  - Japanese Red Cross Osaka Hospital /ID# 207123, Osaka, Osaka
  - Kinki University Sakai Hospital /ID# 166908, Sakai-shi, Osaka
  - The University of Osaka Hospital /ID# 161764, Suita-shi, Osaka
  - Saitama Rihabilitation Center /ID# 168356, Ageo-shi, Saitama
  - Jichi Medical University Saitama Medical Center /ID# 207181, Saitama-shi, Saitama
  - Kamiya Clinic /ID# 261328, Soka-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 212306, Ōtsu, Shiga
  - NHO Matsue Medical Center /ID# 164135, Matsue, Shimane
  - Nanpuh Hospital /ID# 207128, Fujieda-shi, Shizuoka
  - Seirei Hamamatsu General Hospital /ID# 212266, Hamamatsu, Shizuoka
  - Juntendo University Shizuoka Hospital /ID# 207133, Izunokuni-shi, Shizuoka
  - Japanese Red Cross Ashikaga Hospital /ID# 210476, Ashikaga-shi, Tochigi
  - Dokkyo Medical University Hospital /ID# 171050, Mibu, Tochigi
  - Moka Chuo Clinic /ID# 213490, Mooka-shi, Tochigi
  - Mino Tanaka Hospital /ID# 212272, Miyoshi-shi, Tokushima
  - Itsuki Hospital /ID# 164138, Tokushima, Tokushima
  - Juntendo University Hospital /ID# 160823, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 204339, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 207118, Bunkyo-ku, Tokyo
  - National Center of Neurology and Psychiatry /ID# 160824, Kodaira-shi, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center /ID# 260157, Koto-ku, Tokyo
  - Mita Hospital /ID# 207210, Minato-ku, Tokyo
  - Nitobe Memorial Nakano General Hospital /ID# 207377, Nakano-ku, Tokyo
  - Toho University Medical Center Omori Hospital /ID# 212271, Ōta-ku, Tokyo
  - Japanese Red Cross Medical Center /ID# 207129, Shibuya-ku, Tokyo
  - Keio University Hospital /ID# 212267, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 204350, Shinjuku-ku, Tokyo
  - Nomura Neuro Sleep Clinic /ID# 213491, Yonago-shi, Tottori
  - Tottori University Hospital /ID# 207124, Yonago-shi, Tottori
  - Shingu Municipal Medical Center /ID# 207131, Shingu-shi, Wakayama
  - Wakayama Medical University Hospital /ID# 160817, Wakayama, Wakayama
  - Nihonkai General Hospital /ID# 207196, Sakata-shi, Yamagata
  - National Hospital Organization Kanmon Medical Center /ID# 207370, Shimonoseki-shi, Yamaguchi
  - Tokuyama Central Hospital /ID# 171049, Shunan-shi, Yamaguchi
  - Yamaguchi University Hospital /ID# 207774, Ube-shi, Yamaguchi
  - NHO Yanai Medical Center /ID# 164137, Yanai-shi, Yamaguchi
  - University of Yamanashi Hospital /ID# 207120, Chuo-shi, Yamanashi
  - Junwakai Memorial Hospital /ID# 164141, Miyazaki
  - Tachikawa Hospital /ID# 207182, Tachikawa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info. — http://rxabbvie.com